CLINICAL TRIAL: NCT03878966
Title: Polymer Free Drug Eluting Stent in Non ST Elevation Acute Coronary Syndrome
Brief Title: Polymer Free Stent in Acute Coronary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Samir Ali Mahfouz, Assistant lecturer of internal medicine ,critical care unit, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: polymer free stent
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: • Our study will be conducted on at least thirty patients with non-ST-segment elevation acute coronary syndromes (NSTE-ACS)-which include ST depression myocardial infarction and unstable angina- who will be subjected to the early invasive strategy . Polymer-free drug eluting stents will be used for these patients instead of the usually used polymer-permanent drug eluting stents .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Invasive Strategy group (Experimental): * Our study will be conducted on at least thirty patients with non-ST-segment elevation acute coronary syndromes (NSTE-ACS)-which include ST depression myocardial infarction and unstable angina- who will be subjected to the early invasive strategy . Polymer-free drug eluting stents will be used for these patients instead of the usually used polymer-permanent drug eluting stents .
  Interventions: Device: Inserting polymer free drug eluting stent in the coronary arteries

INTERVENTIONS:
Device: Inserting polymer free drug eluting stent in the coronary arteries — • Early invasive strategy with percutaneous coronary intervention will be done for the patients presenting with NST ACS who meet the inclusion criteria using Polymer-free drug eluting stents instead of the polymer-permanent drug eluting stents .

SUMMARY:
To evaluate the short term out comes of the polymer free stents in patients presented with non ST elevation acute coronary syndrome (which include ST depression myocardial infarction and unstable angina ) after percutaneous coronary intervention .

DETAILED DESCRIPTION:
One of the treatment options for CAD is a percutaneous coronary intervention through balloon angioplasty or stent insertion . Although the restenosis rate can be reduced by using bare metal stents , the in-stent restenosis (ISR) rate is still high at around 20%-30% .

increased rates of stent thrombosis were reported with first-generation DESs.(5) The high rate of late and very late stent thrombosis is caused by a long duration of drug elution, which can delay endothelial healing and prolong metallic structure exposure to blood vessel .

Conventionally, DES (drug eluting stents ) are coated with permanent polymers that facilitate drug release and remain long after drug elution is complete. These permanent polymers can cause delayed healing, impaired stent strut endothelialization , and a hypersensitivity reaction, which can culminatein ST (stent thrombosis ).

Research has led to the design of the newer DES (drug eluing stents) that have biodegradable polymers, novel coatings, or are completely polymer free. The polymer-free technology has the potential advantage to reduce the inflammatory and prothrombotic risks related to the utilization of polymers .

* Our study will be conducted on at least thirty patients with non-ST-segment elevation acute coronary syndromes (NSTE-ACS)who will be subjected to the early invasive strategy . Polymer-free drug eluting stents will be used for these patients instead of the usually used polymer-permanent drug eluting stents .
* Patients with NST-ACS who will meet the inclusion and exclusion criteria will be subjected to the following during the admission in the ICU :
* History of the patient concerning :
* Analysis of presenting complaint . Past history of previous similar complaints or the coarse of his illness if he is known to have IHD(ischemic heart disease ) before . Risk factors ( Diabetus mellitus , hypertension , smoking ,....) .Any other co-morbidities and therapeutic history .
* Examination will be done with special concern payied for:
* Blood pressure, heart rate, respiratory rate, Jugular Venous Pressure (JVP), cardiac examination and chest auscultation .
* Investigations in the form of:
* Serial 12 lead ECG .
* Laboratory investigations : (Complete Blood Count (CBC) , Prothrombine time and concentration ,Kidney function ,HCV-Ab , HBs-Ag , HIV Ab , Creatine kinase (CK and CK-MB ) and Troponin at admission and 6 hours later ) .
* Imaging:
* Echocardiographic evaluation with certain emphasis on the following parameters (Wall motion abnormalities ,systolic function , diastolic function and cardiac dimensions).
* TIMI (Thrombolysis in Myocardial Infarction ) risk score will be calculated to every patient .
* Each of the following criteria constitutes one point for TIMI scoring :
* Age ≥65 years
* Three or more risk factors for coronary artery disease (CAD) (family history of CAD, hypertension, hypercholesterolemia, diabetes mellitus, tobacco use)
* Known CAD (stenosis >50%)
* Aspirin use in the past 7 days
* Severe angina (≥2 episodes in 24 hours)
* ST deviation ≥0.5 mm
* Elevated cardiac marker level
* Syntax score will be caiculated during PCI .
* Early invasive strategy with percutaneous coronary intervention will be done for these patients using Polymer-free drug eluting stents instead of the polymer-permanent drug eluting stents .
* The patients will be followed for 6 months after the intervention .
* The patients included in the study will be followed up and re-evaluated at one month and six months after the intervention ( by telephon calls and office visits )
* Re-evaluation will include asking about and analysing symptoms of IHD after the PCI , compliance to the medications .
* Examination: Vital signs , JVP , chest and heart examination .
* 12-lead ECG and cardiac enzymes if needed .
* Follow up Echocardiography will be done at six months .
* Patients will be subjected to follow up diagnostic coronary angiography six months of PCI (whenever possible).
* Six months views after the index procedure coronary angiography will be evaluated by quantitative coronary angiography (QCA) with edge detection method used for evaluation of coronary lesion in index and follow up procedures. Minimal luminal diameter (MLD), Reference vessel diameter (RVD), Percent diameter stenosis %DS), Acute Gain, Late loss and Late loss index will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 85 years of both genders presented with NSTE-ACS with TIMI score ( ≥ 3), who will be subjected to early invasive strategy, whose coronary angiography shows de novo coronary artery disease (CAD) with a stenotic lesion ≥ 70 % requiring use of 2 stents or less.

Exclusion Criteria:

* • Patients with NSTEACS who will be subjected to conservative strategy.

  * Patients whose coronary angiography shows CAD with significant lesions not candidate for PCI like target lesion location in the left main stem or multi vessel disease .
  * In-stent restenosis .
  * Stenosis in bypass graft .
  * Raised renal chemistry (serum creatinine > 2 mg/dl) .
  * Known allergy to the contrast media or other medications used during and after percutaneous coronary intervention .
  * Contraindication to antiplatelet (Asprin, Clopidogrel) or heparin therapy e.g. significant external or internal bleeding and active peptic ulcer .
  * Severly impaired LV systolic function (LVEF < 35%).
  * Malignancies or other co-morbid conditions (for example, severe liver, renal, and pancreatic disease) with life expectancy<6 months or that may result in protocol non-compliance .
  * Pregnancy .
  * Previous enrolment in this trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
• Major adverse cardiac events (MACE) | During six months after the intervention .
  * Recurrent angina pectoris, post-infarction angina, new or recurrent myocardial infarction.
  * Target lesion revascularization (TLR).
  * Target vessel revascularization (TVR).
  * Left ventricular dysfunction.
  * Cardiac arrhythmias.
  * Cardiac death.
Mortality rate | Within six months of the intervention
  Mortality rate in patients underwent the intervention

SECONDARY OUTCOMES:
• Instent restenosis | six months after the intervention
  defined as > 50% instent diameter restenosis on the follow up coronary angiogram.